CLINICAL TRIAL: NCT01477918
Title: Prevalence of Metabolic Syndrome in Patients With Schizophrenia in Korea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yeon-Ho Joo, Professor, Asan Medical Center
Other Study IDs: MetS_1005
Record Dates: First submitted 2011-11-20; First posted 2011-11-23 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Schizophrenia; Metabolic Syndrome
Keywords: prevalence; Korea
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to examine the prevalence of the Metabolic syndrome(MetS) in Korean patients with schizophrenia.

Primary objective:

• To investigate the prevalence of the MetS in Korean patients with schizophrenia

Secondary objectives:

• To compare the prevalence of the MetS among 3 groups according to antipsychotics: typical antipsychotic monotherapy group, atypical antipsychotic monotherapy group, 2 or more antipsychotics group (polypharmacy)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia according to DSM-IV-TR
* Age between 18-65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include all patients that met the following criteria:
  1. Diagnosis of schizophrenia according to DSM-IV-TR
  2. Age between 18-65 years
  To obtain the representative results for the prevalence of the MetS in schizophrenic patients stratified age and gender, we plan to evaluate about one thousand patients in twenty nationwide centers.
  1. 20 centers were selected to provide the representative results of prevalence of the MetS
  2. 50 patients in each center were consecutively enrolled
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-12

PRIMARY OUTCOMES:
prevalence of metabolic syndrome (MetS)
  MetS will be diagnosed according to NCEP ATP III with the Asian-Pacific abdominal obesity criterion (≥90 cm in men, ≥85 cm in women)
  3 or more of the following criteria
  1. fasting plasma glucose >= 100 mg/dl or drug use to treat elevated glucose
  2. serum triglyceride (TG) >= 150 mg/dl or drug use to treat elevated TG
  3. HDL cholesterol level < 40mg /dl in males, < 50 mg/dl in female or drug use to treat low HDL
  4. Systolic BP >=130 mmHg, diastolic BP >=85 or drug use to treat hypertension
  5. Abdominal obesity : above described

CONTACTS AND LOCATIONS:
Locations (1):
- Asan medical center, Seoul, South Korea